CLINICAL TRIAL: NCT05392972
Title: Stress of Anesthesia Professionals in the Operating Room
Acronym: StressBloc
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 00010254 - 2022 - 055
Record Dates: First submitted 2022-05-16; First posted 2022-05-26 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Stress
Keywords: Stress; Professional Resilience; Anaesthesiology; sleep quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Assessment of stress, resilience and associated factors in anesthesia professionals — Assessment of stress, resilience and associated factors in anesthesia professionals

SUMMARY:
The objective of this study was to determine whether there was an association between the resilience of anesthesia professionals in the operating room of the Grenoble University Hospital and perceived work-related stress.

DETAILED DESCRIPTION:
This trial will be conducted at the Grenoble Alpes University Hospital (CHUGA). Volunteer anesthesiologists, anesthesia interns, nurse anesthetists and nurse anesthetist students will answer questionnaires evaluating resilience, perceived stress in the last month, sleep quality, number of hours worked in the month, number of night hours and will evaluate each working day the perceived stress with the visual analogical scale of stress over 3 periods of the working day

The main objective is to determine if there is an association between the resilience (questionnaire: Connord davidson resielience scale: CDRISC10) of the anesthesia professionals in the block of the CHUGA and the perceived stress at work (Perceived stress sacle 10: PSS10).

The secondary objectives are to study the association between:

1. The mean of the two stress VAS (at the beginning and end of the shift) collected and the PSS10 over the same period.
2. The median of the peaks of stress VAS collected and the PSS10 over the same period.
3. The PSS10 and the PSQI (Pittsburgh Sleep Quality Index)
4. The PSS10 and the number of hours worked in the month.
5. The PSS10 and the number of night hours worked in the month.

ELIGIBILITY:
Inclusion Criteria:

* resident in anaesthesiology, Anesthesiologist,anaesthetic nursing student, anaesthetic nurse graduated

Criteria for non-inclusion:

* Professionals objecting to the use of their data in the the research
* Professionals working part-time
* Professionals who had a number of CA > 3 during the month of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: resident in anesthesiology, anesthesiologist, student nurse in anesthesia, volunteer nurse in anesthesia and working at the university hospital center grenoble alpes
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Resilience | at day 0
  Measurement of resilience by Connor-Davidson Resilience Scale 10 (CD RISC 10 from 0 to 40) in participants. A high score indicates better resilience.
Perceived Stress Scale | at day 30
  The Perceived Stress Scale (PSS10 from 10 To 50) measures the degree to which respondents feel their lives are unpredictable, uncontrollable, and overloaded. A high score indicates more stress.

SECONDARY OUTCOMES:
Self-reported stress at the beginning of the workday. | Each work day at the start of the shift. From day 0 to day 30.
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Self-reported stress at the end of the workday. | Every working day at the end of the shift. From day 0 to day 30.
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
Maximum self-reported stress of the workday. | Every working day at the end of the shift. From day 0 to day 30.
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).
The score of the Pittsburgh Sleep Quality Index (PSQI) | at day 30
  The PSQI contains 19 self-assessed questions. These 19 questions combine to yield 7 components: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbance, (6) use of sleeping medication, and (7) daytime dysfunction. Each component gives a score from 0 to 3 points (0 indicates no difficulty, while 3 indicates major difficulty). The scores of the seven components are then added together to give an overall score of 0 to 21 points (0 indicating no difficulty, and 21 indicating major difficulty).
number of hours worked | Each work day at the end of the service. From day 0 to day 30.
  number of hours worked during the working day
number of hours worked at night | Each night of work at the end of the service. From day 0 to day 30.
  the number of hours worked during the work night

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Zafiriou, Principal Investigator — University Hospital, Grenoble; Julien Picard, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France